CLINICAL TRIAL: NCT01423786
Title: Early Oral Nutrition in Mild Acute Pediatric Pancreatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr. Kumar left Nationwide Children's Hospital. The study expired with the Nationwide Children's Hospital on 7/16/14.
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB11-00446; 277711 (Other Grant/Funding Number: The Research Institute at Nationwide Children's Hospital)
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2011-08

CONDITIONS: Acute Pediatric Pancreatitis

ARMS (1):
- Please help (Other): Dr. Kumar left Nationwide Children's Hospital in 2014 and efforts to get ahold of her to complete her ct.gov entries have been unsuccessful as we are not able to get ahold of her.
  In July 2014, she wrote in her Continuing Review application to the NCH IRB: "34 patients have been recruited and data has mostly been collected. Follow up calls have been made and no adverse events occurred during the study period."
  No other information is available.
  Interventions: Dietary Supplement: Early Oral Nutrition

INTERVENTIONS:
Dietary Supplement: Early Oral Nutrition — Once enrolled in the study, patients will be allowed a oral diet that is low in fat.

SUMMARY:
This is a prospective trial for children with the diagnosis of mild acute pancreatitis admitted to the hospital for continued management. Patients will be enrolled in the study within 24 hours of admission/diagnosis and will be allowed an oral diet once enrolled. Demographic, laboratory and imaging data done as standard of care will be collected and additional blood work will be sent as part of the study. Patients will be followed prospectively with regards to tolerance to oral nutrition, pain, length of stay and complications. The hypothesis is that patients that are able to tolerate early oral nutrition will have shorter length of stays and will be similar in terms of pain score ratings, readmission rates, complications and the need for invasive supplemental nutrition. Also patients that are able to tolerate early oral nutrition will have less significant elevation of biochemical markers of pancreatitis severity when compared to patients that do not tolerate early oral nutrition and historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute pancreatitis
* Enroll within 24 hours of diagnosis
* At least 50% of baseline diet must be taken orally

Exclusion Criteria:

* Evidence of severe pancreatitis
* Diagnosis of chronic pancreatitis
* Patients unable to communicate pain or a desire to eat/drink

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-07-16 (Actual); Study Completion 2014-07-16 (Actual)

PRIMARY OUTCOMES:
Tolerance of Oral Nutrition | 1 week
  The time it takes for the patient to tolerate at least 50% of his/her goal oral calories while maintaining hydration as assessed by urine ouput or fluid intake

SECONDARY OUTCOMES:
Length of Stay | 1 week
  The length of time between admission for acute pancreatitis and discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Ellery KM, Kumar S, Crandall W, Gariepy C. The Benefits of Early Oral Nutrition in Mild Acute Pancreatitis. J Pediatr. 2017 Dec;191:164-169. doi: 10.1016/j.jpeds.2017.08.032. Epub 2017 Oct 12. PMID 29031861